CLINICAL TRIAL: NCT00504192
Title: A Phase II Study of Gemcitabine in Combination With Oxaliplatin as First Line Chemotherapy in Patients With Inoperable Biliary Tract Adenocarcinoma
Brief Title: A Phase II Study of Gemcitabine With Oxaliplatin as First Line Chemotherapy in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Dae Sik Hong, Soonchunhyang Bucheon Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH-GO-BTC1
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Advanced Biliary Tract Adenocarcinoma; Gemcitabine; Oxaliplatin; Combination Chemotherapy; Efficacy
MeSH Terms: interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine and Oxaliplatin — gemcitabine 1000mg/m2 IV on day 1 and oxaliplatin 85mg/m2 on day 2 every 2weeks

SUMMARY:
The role of systemic chemotherapy in advanced biliary tract cancer (BTC) is known to be very limited although various single-agent or combination therapies had been tested. However, there is a possibility that palliative chemotherapy induce prolong survival and improve quality of life in advanced BTC based on several studies. A GERCOR study showed the promising result of gemcitabine in combination with oxaliplatin as first line chemotherapy in advanced BTC. Therefore, this phase II trial was planned to investigate efficacy and toxicity of combination chemotherapy with gemcitabine and dose adjusted oxaliplatin in patients with inoperable BTC in Korea.

DETAILED DESCRIPTION:
Treatment scheme

:Gemcitabine 1000 mg/m2/d IV D1 as a 10mg/m2/min Oxaliplatin 85 mg/m2/d IV D2 as a 2 hours infusion

Each cycle is repeated every 2 weeks.

Repeated cycles of treatment will be given for this study unless there is confirmed disease progression or unacceptable toxicity. Subjects will be treated for at least 4 cycles unless there is documented disease progression, unacceptable adverse events or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed biliary tract adenocarcinoma
2. Inoperable disease as defined by:

   * Localized disease in a portion of the liver that does not allow the possibility of complete surgical removal of the tumor with a clear resection margin.

     * Presence of metastatic lesion

       * Unresectable recurrent tumor after curative resection

         * anatomically resectable but inoperable associated with medical condition
3. Biliary obstruction controlled
4. Minimum life expectancy of 12 weeks.
5. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) or evaluable lesion present by imaging study
6. Age over 18 years
7. ECOG performance status of * 2.
8. Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤3xUNL; AST and/or ALT < 5x UNL; Creatinine< 1.5mg/dl or creatinine clearance >50 ml/mins
9. Consent form signed and dated prior to study specific procedures.
10. Subject able to comply with the scheduled follow-up and with the management of toxicities.

Exclusion Criteria:

1. Decompensated Cirrhosis or stage C (Index > 10) according to the Child-Pugh Classification
2. Prior systemic chemotherapy
3. Subject with reproductive potential (M/F) not using adequate contraceptive measures.
4. Pregnancy and breast-feeding.
5. Other serious illness or medical condition, notably heart or lung failure, active uncontrolled infection (infection requiring antibiotics).
6. Past or concurrent history of other neoplasm, except curatively treated basal cell skin cancer or adequately treated in-situ carcinoma of the cervix.
7. Symptomatic or uncontrolled brain metastasis
8. Other concomitant anticancer agent, including Tamoxifen and Interferon.
9. Subjects who cannot be regularly followed up for psychological, social, familial or geographic reasons.
10. Participation in another clinical study or within 30 days before inclusion.
11. History of severe hypersensitivity reactions to gemcitabine or oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
1) To estimate the overall response rate after treatment with gemcitabine and oxaliplatin in patients with advanced biliary tract adenocarcinoma | every 4 cycles

SECONDARY OUTCOMES:
1) To evaluate the safety and tolerability of the treatment combination. 2) To estimate the time to progression and the duration of overall response. 3) To estimate overall tumor growth control rate (CR, PR plus SD). 4) To estimate overall survival. | Overall survival is defined from the first day of treatment to the date of death. Time to progression is defined from the first day of treatment to the date of tumor progression assessed by CT scan or MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Sik Hong, professor, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Kyunggi, South Korea